CLINICAL TRIAL: NCT03633201
Title: Anatomic Congruent Prosthetic Knee Design - a Kinematic and Kinetic Comparison With a Standard Prosthetic Knee Design and the Native Knee
Brief Title: Anatomic Congruent Prosthetic Knee Design
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Regional Hospital Holstebro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: hev-knee-persona001
Record Dates: First submitted 2018-01-18; First posted 2018-08-16 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cruciate Retaining (Active Comparator)
  Interventions: Device: Cruciate Retaining
- Medial Congruent (Active Comparator)
  Interventions: Device: Medial Congruent
- Healthy Controls (No Intervention)

INTERVENTIONS:
Device: Cruciate Retaining — Zimmer Biomet's Personalized Knee system for knee osteoarthritis treatment. The standard insert.
  Other Names: Persona Cruciate Retaining
  Arms: Cruciate Retaining
Device: Medial Congruent — Zimmer Biomet's Personalized Knee system for knee osteoarthritis treatment. The new anatomical congruent shaped insert.
  Other Names: Persona Medial Congruent
  Arms: Medial Congruent

SUMMARY:
This double-blinded randomized control study will use kinematic and kinetic measures to compare an anatomical congruent prosthetic knee design to a standard prosthetic knee design. The patients will be measured pre- and post-operative and compared to a healthy non-osteoarthritis control group.

ELIGIBILITY:
Inclusion Criteria:

* Informed and written consent.
* Primary knee osteoarthritis in capable men and women.
* Indication for cruciate-retaining total knee arthroplasty.

Exclusion Criteria:

* Patients who do not speak and read Danish.
* Patients who are pregnant or at risk of becoming pregnant during the project.
* Patients with active cancer and/or radiation or chemotherapy.
* Patients who are alcoholics or have some form of abuse that impede information and follow-up.
* Patients with severe psychiatric disease that might complicate compliance with follow-up.
* Patients with surgically implants in the affected leg and/or pace maker.
* Patients with greater thigh circumference then 60 cm.
* Patients cannot perform the described exercises.
* Patients with knee instability due to multiligament injury.
* Patients with conditions that severely compromise their gait other than knee osteoarthritis in the affected knee.
* Patients with severe fracture sequelae or severe malalignment at knee level.
* Patients with osteosynthesised fractures using bone graft at knee level.
* Patients with need of an augmentation and/or stem-elongation.
* Patients with metabolic bone disease.
* Patients with rheumatoid arthritis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-07-11 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Kinematics - knee joint movement | 1 year follow-up
  Relative movement (position in millimetres and orientation in degrees) of the knee joint.

SECONDARY OUTCOMES:
Articular joint contact | 1 year follow-up
  Contact between femur and tibia
Kinetic - knee joint contact force | 1 year follow-up
  Internal knee forces (normal and share) of the femur and tibia
Implant inducible micromotion | 1 year follow-up
  Quantifying dynamic inducible micromotion during daily activities.
Static implant migration | 3, 12 and 24 month post operation using first operative day as baseline.
  baseline, three month after surgery and one year after surgery.
Patient Reported Output Measure | 1 year follow-up
  Measured pre- and post operation

CONTACTS AND LOCATIONS:
Overall Officials: Maiken T Stilling, maiken.stilling@clin.au.dk, Principal Investigator — University clinic for hand, hip and knee surgery, Regional Hospital Holstebro, Aarhus University
Locations (1):
- University Clinic of Hand, Hip and Knee Surgery, Regional Hospital Holstebro, Holstebro, Denmark

IPD SHARING:
Plan to Share IPD: No